CLINICAL TRIAL: NCT02726529
Title: Brighter Bites - Access, Continuity and Education With Fruits and Vegetables
Acronym: Brighter Bites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Shreela V Sharma, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-12-0480
Record Dates: First submitted 2016-03-24; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brighter Bites (Experimental): Children of families in the intervention group will also receive the Coordinated Approach to Child Health (CATCH) school-based curriculum in addition to families receiving fresh fruits and vegetables to take home from school once a week along with nutrition education for 8 weeks in Fall and 8 weeks in Spring semesters of the school year.
  Interventions: Behavioral: Brighter Bites; Behavioral: CATCH
- Comparison (Active Comparator)
  Interventions: Behavioral: CATCH

INTERVENTIONS:
Behavioral: Brighter Bites
  Arms: Brighter Bites
Behavioral: CATCH — The comparison schools received training in implementing the Coordinated Approach to Child Health (CATCH) school-based health promotion program

SUMMARY:
The purpose of the research is to find out how well a new nutrition program works for elementary school students and their families. This program is called Brighter Bites. Brighter Bites is a school-based program that teaches students and their parents about the importance of eating fresh fruits and vegetables and how to prepare them in tasty, healthy ways. This project is being carried out at six elementary schools in Houston, Texas. Up to 600 first grade students and their parents/guardians are expected to join this project.

ELIGIBILITY:
Inclusion Criteria:

* Child is in enrolled in the 1st grade in the participating school

Exclusion Criteria:

* None

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 710 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
change intake of servings of fruits and vegetables for the child as assessed using the parent-reported food frequency questionnaire | baseline to 16 weeks
  Child dietary intake was measured using the parent-reported Block Kids Food validated screener to assess children's intake by food group, with outcomes measured in number of servings. The focus of this tool is on intake of fruit and fruit juices, vegetables, potatoes (including French fries), whole grains, meat/poultry/fish, dairy, legumes, saturated fat, "added sugars" (in sweetened cereals, soft drinks, and sweets). A secondary analysis produces estimates for intake of sugary beverages (both kcal and frequency). Individual portion sizes are asked. This screener takes about 10-12 minutes to complete. Servings of fruits and vegetables consumed are cumulatively reported.

SECONDARY OUTCOMES:
change in intake of grams of sugar for the child as assessed using the parent-reported food frequency questionnaire | baseline to 16 weeks
  Child dietary intake was measured using the parent-reported Block Kids Food validated screener to assess children's intake by food group, with outcomes measured in number of servings. The focus of this tool is on intake of fruit and fruit juices, vegetables, potatoes (including French fries), whole grains, meat/poultry/fish, dairy, legumes, saturated fat, "added sugars" (in sweetened cereals, soft drinks, and sweets). A secondary analysis produces estimates for intake of sugary beverages (both kcal and frequency). Individual portion sizes are asked. This screener takes about 10-12 minutes to complete.
change in intake of grams of fat for the child as assessed using the parent-reported food frequency questionnaire | baseline to 16 weeks
  Child dietary intake was measured using the parent-reported Block Kids Food validated screener to assess children's intake by food group, with outcomes measured in number of servings. The focus of this tool is on intake of fruit and fruit juices, vegetables, potatoes (including French fries), whole grains, meat/poultry/fish, dairy, legumes, saturated fat, "added sugars" (in sweetened cereals, soft drinks, and sweets). A secondary analysis produces estimates for intake of sugary beverages (both kcal and frequency). Individual portion sizes are asked. This screener takes about 10-12 minutes to complete.
change in intake of servings of fruits and vegetables for the parent as assessed using the parent-reported food frequency questionnaire | baseline to 16 weeks
  The validated 10-item Fruits and Vegetables Screener by the National Institutes of Health was administered to parents to determine the total number of servings of fruits and vegetables consumed daily.
change in availability of fruits and vegetables in the home as assessed using parent-reported surveys | baseline to 16 weeks
  Parents completed a self-report survey measuring frequency of availability of fresh fruits and vegetables at meals and snacks at home during the past 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Shreela Sharma, PhD, RD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No